CLINICAL TRIAL: NCT04024176
Title: Study of the Parameters of Quantified Gait Analysis in Moderate Hemophiliac Patients (AQM-Hemophile)
Brief Title: Gait Analysis in Moderate Hemophiliac Patients (AQM-Hemophile)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC18_0271
Record Dates: First submitted 2019-05-07; First posted 2019-07-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Moderate Hemophilia; Arthropathy
MeSH Terms: conditions — Joint Diseases | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Each participant will perform the quantified gait analysis examination and a clinical examination. The experiments will be carried out in a single measurement session, including several steps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate hemophiliac patients (Experimental): Each participant will perform a gait analysis and clinical examination
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — The duration of participation of each subject is equal to the duration of the examination, i.e. approximately 30 minutes for the gait analysis and 30 minutes for the clinical examination (including 10 minutes for completing the questionnaire). The experiments will be carried out in a single measurement session, including several steps.

SUMMARY:
The management of moderate hemophilia is less codified than those of severe patients; because these patients are theoretically less likely to bleed and therefore less likely to develop arthropathies. Nowaways, the question arises as to the appropriateness of this "symptomatic" management for the prevention of the occurrence of hemophilic arthropathies. Indeed, a significant number of moderate hemophiliacs seems to develop severe arthropathies that cause significant disability. However, because of the very small proportion of these patients in the total number of hemophiliacs, data are lacking on the impact of arthropathies on this population. The investigators therefore propose to include moderate hemophiliac patients in the study to carry out an evaluation of gait, using a gait analysis to determine the consequences of arthropathies, even sub-clinical ones, according to the duration of the disease's progression. In an associated way, the analysis of different clinical (joint assessment; quality of life score;...), radiological (radiographic; ultrasound (synovial thickness)), biological (level of associated factors ; other associated marker), in order to provide a complete picture of the articular situation in these patients with moderate haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate Hemophilia A or B.
* Have understood the protocol and signed its consent to participate.
* Patient able to perform a walking test.
* Patient affiliated to a social security system

Exclusion Criteria:

* Pregnant women
* Minor
* Majors under guardianship or curatorship
* Refusal to participate;
* Amputee of a lower limb
* Need for technical walking assistance (walking sticks, walker,...).
* Extensive dermatitis of the lower limbs (need for sensor installation for gait analysis);
* Known NYHA (New York Heart Association) grade III or IV heart failure (resting dyspnea);
* Unstable angina or myocardial infarction within three months of inclusion
* Known severe respiratory disease;
* Parkinson's disease, hemiplegia or paraplegia
* Patient unable to understand the objectives or instructions of the study
* Intercurrent pathology likely to modify walking abilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Analysis of spatio-temporal parameters of the gait in moderate hemophiliac patients according to the duration of disease : | during gait analysis and clinical examination (1 hour)
  Analysis of gait parameters
Analysis of kinematic datas of the gait in moderate hemophiliac patients according to the duration of disease : | during gait analysis and clinical examination (1 hour)
  motion capture by optoelectronic system: articular amplitudes at different walking times
Analysis of dynamic datas of the gait in moderate hemophiliac patients according to the duration of disease : | during gait analysis and clinical examination (1 hour)
  accelerations measured by the force platforms during the passage of the subject: moments of force at the different joints during the different walking times

SECONDARY OUTCOMES:
Calculation of the Gait profile Score (GPS) | during gait analysis and clinical examination (1 hour)
  As the Gait Profile Score represents the difference between the patient's data and the average from the reference dataset, the higher the Gait Profile Score value is, the less physiological gait pattern is.
Assessment of joint pain | during gait analysis and clinical examination (1 hour)
  pain (anlog visual scale from 0 (no pain) to 10 (maximal pain))
Assessment of joint health | during gait analysis and clinical examination (1 hour)
  Hemophilia Joint Health score (from 0 (best score) to 25 (worse score))
X-rays of target joints | during gait analysis and clinical examination (1 hour)
  Evaluated by Pettersson's score for hips, knees and ankles (score from 0 (normal score) to 10 (worse score))
Look for synovial hypertrophy by measuring the variation in synovial thickness of the ankles and knees | during gait analysis and clinical examination (1 hour)
  Ultrasound of knees and ankles
evaluation of bleeding and possible increase in synovial angiogenesis | during gait analysis and clinical examination (1 hour)
  Measure of doppler activity

CONTACTS AND LOCATIONS:
Overall Officials: Alban Fouasson Chailloux, Dr, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Department of Physical Medicine and Locomotive Rehabilitation (Nantes University Hospital), Nantes
  - Department of Physical Medicine and Neurological Rehabilitation (Nantes University Hospital), Nantes
  - Regional Hemophilia Treatment Centre (Nantes University Hospital), Nantes
  - Rheumatology department (Nantes University Hospital), Nantes